CLINICAL TRIAL: NCT02638844
Title: ARDStrain : Assessment of Right Ventricular 2d-strain in Acute Respiratory Distress Syndrome
Brief Title: Assessment of Right Ventricular 2d-strain in Acute Respiratory Distress Syndrome
Acronym: ARDStrain
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Other Study IDs: CPRC2013 ARDStrain
Record Dates: First submitted 2015-12-16; First posted 2015-12-23 (Estimated); Last update posted 2018-02-05 (Actual); Status verified 2017-07

CONDITIONS: ARDS
Keywords: echocardiography

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Assessment of right ventricular (RV) function in patients with acute respiratory syndrome (ARDS) is warranted because RV failure is frequent and associated with worse outcome. Transthoracic echocardiography is the cornerstone of RV assessment but it remains challenging. Quantification of RV deformation by speckle-tracking imaging echocardiography (STE) is a widely available and reproducible technique that readily provides an integrated analysis of all segments of the RV. This study aims to investigate the accuracy of STE-derived strain parameters in assessing RV function during ARDS.

ELIGIBILITY:
Inclusion Criteria:

* patients with moderate or severe ARDS (Berlin definition)
* receiving mechanical ventilation (>48h estimated length)
* Transthoracic echocardiography performed during the first 36h after ICU admission

Exclusion Criteria:

* pregnancy
* protected or deprived of Liberty major
* chronic respiratory disease
* history of clinical right heart failure
* chronic heart failure with LVEF < 35%
* severe valvular heart disease
* under 18 or protected-adults

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ICU patients with moderate or severe ARDS receiving invasive mechanical ventilation
Sampling Method: Non-Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2015-12; Primary Completion 2017-07 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Measure of longitudinal peak systolic strain | up to 36 hours after Intensive Care Unit admission

SECONDARY OUTCOMES:
Measure of PaO2/FiO2 ratio | up to 36 hours after Intensive Care Unit admission
Ventilator-free days | 28 days
Mortality | 28 days

CONTACTS AND LOCATIONS:
Locations (1):
- Lemarie Jeremie, Nancy, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lemarie J, Maigrat CH, Kimmoun A, Dumont N, Bollaert PE, Selton-Suty C, Gibot S, Huttin O. Feasibility, reproducibility and diagnostic usefulness of right ventricular strain by 2-dimensional speckle-tracking echocardiography in ARDS patients: the ARD strain study. Ann Intensive Care. 2020 Feb 13;10(1):24. doi: 10.1186/s13613-020-0636-2. PMID 32056017